CLINICAL TRIAL: NCT05832385
Title: Effects of Different Radiation Dosimetry for Anorectal Function of Patients With Pelvic Cancer: a Study Protocol for a Prospective, Observational, Controlled, Multicenter Study
Brief Title: Effects of Different Radiation Dosimetry for Anorectal Function of Patients With Pelvic Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hongcheng Lin, vice chief of department of anus and intestine surgery, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2023ZSLYEC-039
Record Dates: First submitted 2023-02-14; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Anorectal Cancer
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- radiation dose≤50Gy: rectal cancer with IMRT radiation dose≤50Gy
- radiation dose>50Gy: anal cancer with IMRT radiation dose>50Gy
  Interventions: Radiation: IMRT

INTERVENTIONS:
Radiation: IMRT — anal cancer: chemoradiotherapy, radiation dose>50Gy; rectal cancer: chemoradiotheray, radiation dose=50Gy
  Other Names: chemotherapy
  Groups: radiation dose>50Gy

SUMMARY:
In this prospective, open, multicenter, multi-arm, observational controlled study, the investigators investigated the impact of different pelvic radiation doses of anal cancer and rectal cancer patients on the dynamic changes of anal function, and analyzed the correlation between the changes of anal function and the score of anal incontinence in the radiation dose≤50Gy group and >50Gy group. The study population includes 124 patients with anal canal cancer or rectal cancer who have received sphincter preservation treatments (including radiochemotherapy), aged from 18 to 75 years old undergoing sphincter preservation treatments at The Sixth Affiliated Hospital, Sun Yat-sen University and Nanfang Hospital, Southern Medical University. The primary outcome is the average resting pressure of anal sphincter. The secondary outcomes are maximum anal sphincter contraction pressure and Wexner continence score. Evaluations will be carried out at the following stages: baseline (T1), after radiotherapy or chemotherapy (before surgery, T2), after surgery (before closing the temporary stoma, T3), and at follow-up visits (every 3 to 6 months, T4, T5……). Follow-up for each patient will be at least 2 years.

ELIGIBILITY:
Inclusion criteria 18-75 years of age. Anal cancer and rectal cancer with pathological diagnosis. Patient will undergo sphincter-preserving therapies. Eastern Cooperative Oncology Group (ECOG) score for performance status is 0-2. Written informed consent. Exclusion criteria Patients who have undergone pelvic surgery, such as rectal cancer surgery and gynaecological procedures. Patients who have received pelvic radiotherapy. Patients with other active malignant tumors. Patients with a history of prior peri-anal abscess, anorectal trauma, and inflammatory bowel disease (IBD).

Recently (less than 4 weeks) received surgery or patients with recent severe trauma.

Significant cardiac disease: congestive heart failure of New York Heart Association class ≥2; patients with recent (less than 12 months) active coronary artery disease (unstable angina or myocardial infarction).

Recent (less than 6 months) thrombosis or embolism events, such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism and deep vein thrombosis.

Patients with toxicity (Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥ 2) caused by previous treatment that has not subsided.

Women who suffered anal sphincter tear after vaginal delivery. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with anal and rectal cancer at The Sixth Affiliated Hospital, Sun Yat-sen University and Nanfang Hospital, Southern Medical University will be assessed for suitability for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
the average resting pressure of anal sphincter | 2023.05-2026.05
  High-resolution anorectal manometry will be used to assess the average resting pressure and maximal contraction pressure.

SECONDARY OUTCOMES:
maximum anal sphincter contraction pressure | 2023.05-2026.05
  High-resolution anorectal manometry will be used to assess the average resting pressure and maximal contraction pressure.
Wexner continence score | 2023.05-2026.05
  Wexner continence score 0-20, higher means worse